CLINICAL TRIAL: NCT05098639
Title: An Adaptive Mobile Intervention to Increase Safe Drinking Strategies Using Deviance Regulation Theory
Brief Title: DRT Mobile Intervention to Increase Safe Drinking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001422
Record Dates: First submitted 2021-09-10; First posted 2021-10-28 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Alcohol; Use, Problem
Keywords: Alcohol Use; Deviance Regulation Theory; Mobile Intervention; Protective Behavioral Strategies
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: This study will randomly assign participants to one of three conditions: Active Control (BASICS), DRT, or DRT+Active Control
Who Masked: Participant
Masking Description: Participants will be unaware of the condition they are in. As the initial session requires a brief individual session using BASICS, DRT, or DRT+BASICS, investigators will be aware of study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BASICS (Active Comparator): Participants in the active control will receive a modified single session BASICS. BASICS is a well-documented and empirically supported prevention/intervention program for college student drinkers. BASICS targets heavy drinking students that have experienced or are at an increased risk for a variety of alcohol-related problems linked to college student life. The program is designed to help students make better alcohol-use decisions based on a broader understanding of the risks associated with problem drinking. It enhances motivation to change and promotes the development of skills to moderate drinking. The overall style of the program uses motivational interviewing and emphasizes empathy and non-judgmental interaction. The aims of BASICS are to (1) reduce alcohol consumption and consequences, (2) promote healthier and more responsible choices, and (3) provide information and coping skills.
  Interventions: Behavioral: BASICS
- Deviance Regulation Theory (Experimental): DRT participants receive an initial intervention session that is consistent with their current (pre-intervention) PBS frequency norm beliefs. For the initial intervention session, participants discuss their perception of the use of alcohol and use of protective behavioral strategies among campus peers. They are given feedback on the injunctive norms of alcohol use and PBS use by their peers which is tailored to each individuals normative perceptions. Following the initial intervention session, participants will carry a mobile device that allows for individuals to report current drinking environments. They then receive DRT consistent feedback based on the norms reported in their current drinking environment.
  Interventions: Behavioral: Deviance Regulation Theory (DRT)
- Deviance Regulation Theory+BASICS (Experimental): DRT participants receive an initial intervention session that is consistent with their current (pre-intervention) PBS frequency norm beliefs but also follows the framework of BASICS. For the initial intervention session, participants discuss their perception of the use of alcohol and use of protective behavioral strategies among campus peers. They are given feedback on both descriptive and injunctive norms of alcohol use and PBS use by their peers which is tailored to each individuals normative perceptions. Following the initial intervention session, participants will carry a mobile device that allows for individuals to report current drinking environments. They then receive DRT consistent feedback based on the norms reported in their current drinking environment.
  Interventions: Behavioral: BASICS; Behavioral: Deviance Regulation Theory (DRT)

INTERVENTIONS:
Behavioral: BASICS — In the BASICS condition, individuals receive information about alcohol use on campus and discuss safe drinking practices. They also receive personalized normative feedback based on their alcohol use and their use of protective behavioral strategies.
  Arms: BASICS; Deviance Regulation Theory+BASICS
Behavioral: Deviance Regulation Theory (DRT) — The Deviance Regulation Intervention comprises tailored intervention messages based on perceived norms. Participants complete an initial session that focuses on perceived norms of protective behavioral strategy (PBS) use and heavy drinking among peers. The therapist engages participants in a tailored discussion based on their perceived norms. If individuals believe PBS use is uncommon, the therapist discusses the positive social image that PBS use portrays. If the participant believes PBS is common, the therapist engages the participant in discussion of the negative aspects of non-PBS use. A similar strategy is taken for common and uncommon heavy alcohol use. Finally, the participant carries a mobile device which provide real-time adaptive positive or negative messages (consistent with the initial session) based on the perceived drinking and PBS norms of their current drinking environment.
  Arms: Deviance Regulation Theory; Deviance Regulation Theory+BASICS

SUMMARY:
The current project uses a brief mobile intervention, grounded in Deviance Regulation Theory, to deliver in-the-moment messaging meant to increase responsible drinking among college students. Participants receive positive messages about individuals that use responsible drinking behaviors or negative messages about individuals that do not use responsible drinking behaviors. It is hypothesized that these messages delivered at appropriate times will differentially affect use of responsible drinking behaviors as a function of individual beliefs about the prevalence of responsible drinking among peers.

DETAILED DESCRIPTION:
College student alcohol use remains a significant public health issue. College students consume alcohol at higher rates than their non-college peers. Though most college students "mature out" of heavy alcohol use by graduation, the consequences resulting from frequent acute intoxication during college can be devastating. Identifying cost effective ways to reduce problematic alcohol use, that can be widely disseminated, remains vitally important. A large body of literature has examined associations between social norms and drinking among college students. Several college drinking interventions have utilized social norms to reduce alcohol use and alcohol-related consequences. However, recent research suggests these interventions may not be as effective as once though. Despite the support for social norms as an etiological basis for heavy drinking, and its implementation in interventions, the operationalization has remained relatively narrow. Social norms interventions have generally not taken broader theoretical perspectives into account. Nor have they been applied much beyond the exclusive focus on quantity and frequency of consumption. The present study addresses these issues by examining the effects of an intervention grounded in Deviance Regulation Theory, meant to increase use of alcohol protective behavioral strategies when drinking. Deviance Regulation Theory posits that individuals will seek to engage in behaviors that allow them to standout in positive ways or avoid standing-out in negative ways. Both of these effects are based on the perception of the behavioral norm. Participants are randomly assigned to receive messages that presents individuals who DO use PBS in a positive light, information that presents individuals who DO NOT use PBS in a negative light, or an active control (BASICS). It is hypothesized that among individuals who believe PBS use is uncommon among their peers, positive messages about PBS users will result in increased PBS use, and subsequent decreases in alcohol use and problems. In contrast among individuals who believe PBS use is common among their peers, negative messages about PBS users will result in increased PBS use, and subsequent decreases in alcohol use and alcohol problems. If successful this trial will pave the way for a novel intervention for college students that can be tailored to individual beliefs about PBS use norms and that could be combined with existing interventions for college student drinking.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Severe mental illness
* Under 18 years of age
* Over 26 years of age
* Unable to speak English fluently

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Protective Behavioral Strategies- Pre-Intervention | Past three months prior to intervention/study
  Protective behavioral strategies (PBS) are harm-reduction strategies to decrease alcohol-related consequences when consuming alcohol. There are three subtypes: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times). PBS are assessed in this study using the Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use will be reported on a five-point Likert-scale from 0 (Never) to 4 (Always). The mean score across all 20 items serves as the outcome variable. Participants are asked to record their PBS use from the past three months. Scores range from 0 to 20. Higher scores indicate greater use of protective strategies.
Protective Behavioral Strategies- Initial intervention (Week 1) | Past week before intervention
  Protective behavioral strategies (PBS) are harm-reduction strategies to decrease alcohol-related consequences when consuming alcohol. There are three subtypes: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times). PBS are assessed in this study using the Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use will be reported on a five-point Likert-scale from 0 (Never) to 4 (Always). The mean score across all 20 items serves as the outcome variable. Participants are asked to record their PBS use from the past week. Scores range from 0 to 20. Higher scores indicate greater use of protective strategies.
Protective Behavioral Strategies- Week 2 | Past 1 week measured- 1 week post intervention
  Protective behavioral strategies (PBS) are harm-reduction strategies to decrease alcohol-related consequences when consuming alcohol. There are three subtypes: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times). PBS are assessed in this study using the Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use will be reported on a five-point Likert-scale from 0 (Never) to 4 (Always). The mean score across all 20 items serves as the outcome variable. Participants are asked to record their PBS use from the past week. Scores range from 0 to 20. Higher scores indicate greater use of protective strategies.
Protective Behavioral Strategies- Week 3 | Past 1 week measured-2 weeks post intervention
  Protective behavioral strategies (PBS) are harm-reduction strategies to decrease alcohol-related consequences when consuming alcohol. There are three subtypes: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times). PBS are assessed in this study using the Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use will be reported on a five-point Likert-scale from 0 (Never) to 4 (Always). The mean score across all 20 items serves as the outcome variable. Participants are asked to record their PBS use from the past week. Scores range from 0 to 20. Higher scores indicate greater use of protective strategies.
Protective Behavioral Strategies- Week 4 | Past 1 week measured-3 weeks post intervention
  Protective behavioral strategies (PBS) are harm-reduction strategies to decrease alcohol-related consequences when consuming alcohol. There are three subtypes: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times). PBS are assessed in this study using the Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use will be reported on a five-point Likert-scale from 0 (Never) to 4 (Always). The mean score across all 20 items serves as the outcome variable. Participants are asked to record their PBS use from the past week. Scores range from 0 to 20. Higher scores indicate greater use of protective strategies.
Protective Behavioral Strategies- 3 month follow up | Past 3 months measured- 12 week post intervention
  Protective behavioral strategies (PBS) are harm-reduction strategies to decrease alcohol-related consequences when consuming alcohol. There are three subtypes: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times). PBS are assessed in this study using the Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use will be reported on a five-point Likert-scale from 0 (Never) to 4 (Always). The mean score across all 20 items serves as the outcome variable. Participants are asked to record their PBS use from the past three months. Scores range from 0 to 20. Higher scores indicate greater use of protective strategies.
Protective Behavioral Strategies- 6 month follow-up | Past 3 months measured- 26 weeks post intervention
  Protective behavioral strategies (PBS) are harm-reduction strategies to decrease alcohol-related consequences when consuming alcohol. There are three subtypes: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times). PBS are assessed in this study using the Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use will be reported on a five-point Likert-scale from 0 (Never) to 4 (Always). The mean score across all 20 items serves as the outcome variable. Participants are asked to record their PBS use from the past three months. Scores range from 0 to 20. Higher scores indicate greater use of protective strategies.

SECONDARY OUTCOMES:
Alcohol-related consequences- Pre-intervention | Past three months prior to intervention/study
  Alcohol-related consequences are assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants record alcohol consequences (Yes/No/ I do not wish to respond) from the past three months. Scores can range from 0-48. Higher scores indicate a greater number of alcohol consequences.
Alcohol-related consequences- Initial intervention (Week 1) | Past week before intervention
  Alcohol-related consequences are assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants record alcohol consequences (Yes/No/ I do not wish to respond) from the past week. Scores can range from 0-48. Higher scores indicate a greater number of alcohol consequences.
Alcohol-related consequences- Week 2 | Past 1 week measured- 1 week post intervention
  Alcohol-related consequences are assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants record alcohol consequences (Yes/No/ I do not wish to respond) from the past week. Scores can range from 0-48. Higher scores indicate a greater number of alcohol consequences.
Alcohol-related consequences- Week 3 | Past 1 week measured- 2 week post intervention
  Alcohol-related consequences are assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants record alcohol consequences (Yes/No/ I do not wish to respond) from the past week. Scores can range from 0-48. Higher scores indicate a greater number of alcohol consequences.
Alcohol-related consequences- Week 4 | Past 1 week measured- 3 week post intervention
  Alcohol-related consequences are assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants record alcohol consequences (Yes/No/ I do not wish to respond) from the past week. Scores can range from 0-48. Higher scores indicate a greater number of alcohol consequences.
Alcohol-related consequences- 3 month follow up | Past 3 months measured- 12 week post intervention
  Alcohol-related consequences are assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants record alcohol consequences (Yes/No/ I do not wish to respond) from the past week. Scores can range from 0-48. Higher scores indicate a greater number of alcohol consequences.
Alcohol-related consequences- 6 month follow-up | Past 3 months measured- 26 weeks post intervention
  Alcohol-related consequences are assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants record alcohol consequences (Yes/No/ I do not wish to respond) from the past three months. Scores can range from 0-48. Higher scores indicate a greater number of alcohol consequences.
Alcohol use- Pre-intervention | Past three months prior to intervention/study
  Alcohol use (quantity) is assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M uses a grid to report typical number of drinks consumed for an average day in an average week, over the last three months. The DDQ-M is used to measure the number of drinks consumed for each day of the week. These are summed across the days of the week to provide a measure of typical standard drinks consumed. The lower limit is 0, there is no upper limit as this is a self-reported number. Higher numbers indicate more alcohol is consumed.
Alcohol use- Initial intervention (Week 1) | Past week before intervention
  Alcohol use (quantity) is assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M uses a grid to report typical number of drinks consumed for an average day in an average week, over the last week. The DDQ-M is used to measure the number of drinks consumed for each day of the last week. These are summed across the days of the week to provide a measure of standard drinks consumed for the previous week. The lower limit is 0, there is no upper limit as this is a self-reported number. Higher numbers indicate more alcohol is consumed.
Alcohol use- Week 2 | Past 1 week measured- 1 week post intervention
  Alcohol use (quantity) is assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M uses a grid to report typical number of drinks consumed for an average day in an average week, over the last week. The DDQ-M is used to measure the number of drinks consumed for each day of the last week. These are summed across the days of the week to provide a measure of standard drinks consumed for the previous week. The lower limit is 0, there is no upper limit as this is a self-reported number. Higher numbers indicate more alcohol is consumed.
Alcohol use- Week 3 | Past 1 week measured- 2 weeks post intervention
  Alcohol use (quantity) is assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M uses a grid to report typical number of drinks consumed for an average day in an average week, over the last week. The DDQ-M is used to measure the number of drinks consumed for each day of the last week. These are summed across the days of the week to provide a measure of standard drinks consumed for the previous week. The lower limit is 0, there is no upper limit as this is a self-reported number. Higher numbers indicate more alcohol is consumed.
Alcohol use- Week 4 | Past 1 week measured- 3 weeks post intervention
  Alcohol use (quantity) is assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M uses a grid to report typical number of drinks consumed for an average day in an average week, over the last week. The DDQ-M is used to measure the number of drinks consumed for each day of the last week. These are summed across the days of the week to provide a measure of standard drinks consumed for the previous week. The lower limit is 0, there is no upper limit as this is a self-reported number. Higher numbers indicate more alcohol is consumed.
Alcohol use- 3 month follow up | Past 3 months measured- 12 week post intervention
  Alcohol use (quantity) is assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M uses a grid to report typical number of drinks consumed for an average day in an average week, over the last three months. The DDQ-M is used to measure the number of drinks consumed for each day of the week. These are summed across the days of the week to provide a measure of typical standard drinks consumed. The lower limit is 0, there is no upper limit as this is a self-reported number. Higher numbers indicate more alcohol is consumed.
Alcohol use- 6 month follow up | Past 3 months measured- 24 week post intervention
  Alcohol use (quantity) is assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M uses a grid to report typical number of drinks consumed for an average day in an average week, over the last three months. The DDQ-M is used to measure the number of drinks consumed for each day of the week. These are summed across the days of the week to provide a measure of typical standard drinks consumed. The lower limit is 0, there is no upper limit as this is a self-reported number. Higher numbers indicate more alcohol is consumed.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be uploaded to the OSF page for this study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 mo. post data collection
URL: https://osf.io/d6zke/